CLINICAL TRIAL: NCT05438589
Title: Evaluation of the Performance of Novel Rapid Diagnostics for SARS-CoV-2 at Point-of-care
Brief Title: Novel Rapid POC Diagnostics for COVID-19
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CV008
Record Dates: First submitted 2022-06-29; First posted 2022-06-30 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multicentre study in which the diagnostic accuracy of multiple Covid-19 Antigen rapid diagnostic tests will be assessed for COVID-19 case detection using prospectively collected nasal swabs and saliva samples from participants suspected to have Covid-19 infection (with or without symptoms). The study will last approximately 9 months.

DETAILED DESCRIPTION:
Adult individuals with presumptive Covid-19, either symptomatic or asymptomatic, will be screened for inclusion at 4 different study sites located in Georgia and South Africa.

Enrolled participants will be asked to provide 2 samples: one nasopharyngeal swab that will be utilized for Covid-19 diagnosis by standard PCR and one sample (either nasal swab or saliva) to be used for the new antigen rapid diagnostic test under evaluation. At least 2 different antigen tests will be evaluated to determine sensitivity and specificity: Novel Corona Virus (SARS-CoV-2) Ag Rapid Test Kit (Jiangsu Bioperfectus Technologies) and GeneFinder COVID-19 Ag Rapid test (Osang Healthcare).

The data gathered from this study, could be used as part of the dossier to be submitted to WHO (world health organization) for review.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Presenting to testing locations linked to the clinical sites
* Suspected to have COVID-19 (as per WHO or national guidelines). These include the following groups:

  * Individuals with acute onset of any of the following signs or symptoms: fever, cough, general weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnoea, anorexia/nausea/vomiting, diarrhoea, altered mental status (for SYMPTOMATIC group);
  * Contacts of confirmed cases of COVID-19
  * Individuals residing or working in an area with high risk of transmission of virus
  * Individuals residing or travelling to an area with community transmission
  * Individuals working in any health care setting, including within health facilities or within the community
* Provided voluntary written consent to participate in this study
* Provided a specimen suitable for testing

Exclusion Criteria:

* Individuals unable to cooperate with respiratory sample collection
* Individuals on oxygen therapy
* Recent history of excessive nose bleeds
* Individuals unable to give informed consent
* Hemodynamic instability as determined by the treating physician

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals (≥ 18 years old) suspected to have COVID-19 (as per national or WHO guidelines) presenting at the testing site(s) will be invited to participate. Each participant will have two respiratory swabs collected: one for RT-PCR testing and diagnosis, paired with a second swab to be used on the index Ag RDT. In order to meet the study objectives, two different population groups will be considered:
  1. SYMPTOMATIC: Individuals (≥ 18 years old) suspected to have COVID-19 (as per national or WHO guidelines) and presenting at the testing site(s) with symptoms of COVID-19.
  2. ASYMPTOMATIC: Individuals (≥ 18 years old) at risk of COVID-19 (as per national or WHO guidelines) and presenting at the testing site(s) with no symptoms of COVID-19
Sampling Method: Probability Sample
Enrollment: 1283 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | at enrolment
  Point estimates of sensitivity and specificity of index test, with 95% confidence intervals, using RT-PCR as reference standard

SECONDARY OUTCOMES:
Sensitivity and specificity in specific subgroups | at enrolment
  Point estimates of sensitivity and specificity of index test with 95% confidence intervals in specific subgroups defined based on presence of the symptoms, disease stage (days since symptom onset, e.g. acute, early, late), severity of symptoms, RT-PCR Ct values, vaccination status

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ivanova Reipold, MD, PhD, Principal Investigator — Find
Locations (2):
- National Center for Disease Control, Tbilisi, Georgia
- Ezintsha, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided